CLINICAL TRIAL: NCT02230956
Title: BOTOX® Efficacy and Safety in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622-145; 2014-001076-58 (EudraCT Number)
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- OnabotulinumtoxinA 400 U (Experimental): OnabotulinumtoxinA 400 U injection into the intra-articular space of the study knee on Day 1.
  Interventions: Biological: onabotulinumtoxinA
- OnabotulinumtoxinA 200 U (Experimental): OnabotulinumtoxinA 200 U injection into the intra-articular space of the study knee on Day 1.
  Interventions: Biological: onabotulinumtoxinA
- Placebo (Placebo Comparator): Placebo (Normal Saline) injection into the intra-articular space of the study knee on Day 1.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: onabotulinumtoxinA — onabotulinumtoxinA (botulinum toxin Type A) injection into the intra-articular space of the study knee.
  Other Names: botulinum toxin Type A; BOTOX®
  Arms: OnabotulinumtoxinA 200 U; OnabotulinumtoxinA 400 U
Drug: Normal Saline — Normal Saline (placebo) injection into the intra-articular space of the study knee.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of a single intra-articular injection of 2 doses of BOTOX® (onabotulinumtoxinA) compared with placebo as treatment for knee osteoarthritis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Painful osteoarthritis
* Able to discontinue anti-inflammatory drugs and analgesics
* Must be ambulatory without assistive walking devices

Exclusion Criteria:

* Chronic pain conditions other than knee osteoarthritis
* Treatment with corticosteroids in the study knee within 12 weeks
* Treatment with hyaluronic acid in the study knee within 24 weeks
* Previous treatment with any botulinum toxin for any reason
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (3):
- Artesia, California, United States
- Pardubice, Czechia
- Vejle, Denmark

REFERENCES:
- [Derived] McAlindon TE, Schmidt U, Bugarin D, Abrams S, Geib T, DeGryse RE, Kim K, Schnitzer TJ. Efficacy and safety of single-dose onabotulinumtoxinA in the treatment of symptoms of osteoarthritis of the knee: results of a placebo-controlled, double-blind study. Osteoarthritis Cartilage. 2018 Oct;26(10):1291-1299. doi: 10.1016/j.joca.2018.05.001. Epub 2018 May 9. PMID 29753118
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Started | 44 | 43 | 89
Completed | 39 | 37 | 82
Not Completed | 5 | 6 | 7
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Personal Reasons | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Other Miscellaneous Reason | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo | Total
Number analyzed (Participants) | 44 | 43 | 89 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.25) | 60.2 (8.41) | 61.1 (7.79) | 60.8 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 26 | 51 | 107
  Male | 14 | 17 | 38 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 7-Day Average Daily Pain Score Using an 11-Point Scale
Description: Participants recorded the pain in their knee during the previous 24 hours in a daily diary where: 0=no pain to 10= worst pain possible. The daily pain scores over 7-days were averaged. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 8
Population: Safety population consisted of all randomized participants who received the study treatment and were analyzed by treatment actually received.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Number analyzed (Participants) | 44 | 43 | 89
score on a scale
  Baseline | 5.92 (1.222) | 6.09 (1.313) | 6.00 (1.150)
  Change from Baseline at Week 8 | -1.68 (1.641) | -2.07 (1.602) | -1.98 (1.793)

2. Secondary Outcome: Change From Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC™) Pain Score Using an 11-Point Scale
Description: The WOMAC Pain Score consisted of 5 questions about pain completed by the participant where: 0=no pain to 10=extreme pain for a total possible Pain Score of 0 (best) to 50 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 1, 4, 8, 12, 16, 20 and 24
Population: Safety population consisted of all randomized participants who received the study treatment and were analyzed by treatment actually received. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Number analyzed (Participants) | 44 | 43 | 89
score on a scale
  Baseline | 5.84 (1.629) | 5.41 (1.806) | 5.34 (1.548)
  Change from Baseline at Week 1: number analyzed (Participants) | 44 | 43 | 88
  Change from Baseline at Week 1 | -1.75 (1.567) | -1.61 (1.666) | -1.62 (1.805)
  Change from Baseline at Week 4: number analyzed (Participants) | 43 | 43 | 86
  Change from Baseline at Week 4 | -1.82 (1.893) | -1.67 (1.763) | -1.81 (1.848)
  Change from Baseline at Week 8: number analyzed (Participants) | 40 | 39 | 84
  Change from Baseline at Week 8 | -2.02 (1.899) | -1.52 (1.907) | -1.76 (1.976)
  Change from Baseline at Week 12: number analyzed (Participants) | 39 | 39 | 84
  Change from Baseline at Week 12 | -1.81 (1.975) | -1.82 (1.870) | -1.75 (2.014)
  Change from Baseline at Week 16: number analyzed (Participants) | 40 | 38 | 80
  Change from Baseline at Week 16 | -1.67 (1.841) | -1.64 (2.174) | -1.62 (1.901)
  Change from Baseline at Week 20: number analyzed (Participants) | 39 | 38 | 80
  Change from Baseline at Week 20 | -1.79 (1.937) | -1.68 (2.066) | -1.78 (2.037)
  Change from Baseline at Week 24: number analyzed (Participants) | 39 | 37 | 82
  Change from Baseline at Week 24 | -1.93 (2.289) | -1.81 (2.181) | -1.69 (2.008)

3. Secondary Outcome: Change From Baseline in the WOMAC™ Physical Function Score Using an 11-Point Scale
Description: The WOMAC Physical Function Score consisted of 17 questions about the difficulty of daily activities completed by the participant where: 0=no difficulty to 10=extreme difficulty for a total possible Physical Function Score of 0 (best) to 170 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 1, 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Number analyzed (Participants) | 44 | 43 | 89
score on a scale
  Baseline | 5.56 (1.804) | 5.35 (1.995) | 4.99 (1.854)
  Change from Baseline at Week 1: number analyzed (Participants) | 44 | 43 | 88
  Change from Baseline at Week 1 | -1.33 (1.424) | -1.64 (1.870) | -1.44 (1.933)
  Change from Baseline at Week 4: number analyzed (Participants) | 43 | 43 | 86
  Change from Baseline at Week 4 | -1.26 (1.672) | -1.66 (1.908) | -1.35 (2.069)
  Change from Baseline at Week 8: number analyzed (Participants) | 40 | 39 | 84
  Change from Baseline at Week 8 | -1.54 (1.819) | -1.50 (2.043) | -1.27 (2.070)
  Change from Baseline at Week 12: number analyzed (Participants) | 39 | 39 | 84
  Change from Baseline at Week 12 | -1.30 (1.648) | -1.68 (1.781) | -1.40 (2.170)
  Change from Baseline at Week 16: number analyzed (Participants) | 40 | 38 | 80
  Change from Baseline at Week 16 | -1.29 (1.558) | -1.59 (2.127) | -1.09 (1.991)
  Change from Baseline at Week 20: number analyzed (Participants) | 39 | 38 | 80
  Change from Baseline at Week 20 | -1.34 (1.651) | -1.44 (2.172) | -1.18 (2.087)
  Change from Baseline at Week 24: number analyzed (Participants) | 39 | 37 | 82
  Change from Baseline at Week 24 | -1.48 (2.029) | -1.56 (2.232) | -1.12 (1.998)

4. Secondary Outcome: Patient Global Impression of Change (GIC) Using a 7-Point Scale
Description: The participant rated the change in their health status since enrollment using a 7-point scale where: +3=very much improved, +2=much improved, +1=minimally improved, 0=no change, -1=minimally worse, -2=much worse and -3=very much worse. Negative scores indicate worsening and positive scores indicate improvement.
Time Frame: Weeks 1, 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Number analyzed (Participants) | 44 | 43 | 89
score on a scale
  Week 1: number analyzed (Participants) | 44 | 43 | 87
  Week 1 | 0.9 (1.00) | 1.2 (0.97) | 1.1 (1.09)
  Week 4: number analyzed (Participants) | 43 | 43 | 86
  Week 4 | 0.9 (1.24) | 1.2 (1.23) | 1.2 (1.10)
  Week 8: number analyzed (Participants) | 40 | 39 | 84
  Week 8 | 1.1 (1.09) | 0.9 (1.35) | 1.0 (1.00)
  Week 12: number analyzed (Participants) | 39 | 39 | 84
  Week 12 | 1.1 (1.35) | 1.2 (1.30) | 1.0 (1.14)
  Week 16: number analyzed (Participants) | 40 | 38 | 80
  Week 16 | 1.1 (1.31) | 1.1 (1.36) | 1.0 (1.10)
  Week 20: number analyzed (Participants) | 39 | 38 | 80
  Week 20 | 1.1 (1.24) | 1.0 (1.42) | 1.0 (1.20)
  Week 24: number analyzed (Participants) | 39 | 37 | 82
  Week 24 | 0.8 (1.34) | 1.0 (1.41) | 0.9 (1.28)

5. Secondary Outcome: Change From Baseline in the 7-Day Average Daily Worst Pain Score Using an 11-Point Scale
Description: Participants recorded the pain in their knee during the previous 24 hours in a daily diary where: 0=no pain to 10= worst pain possible. The daily worst pain scores over 7-days were averaged. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Number analyzed (Participants) | 44 | 43 | 89
score on a scale
  Baseline | 6.50 (1.243) | 6.84 (1.342) | 6.63 (1.157)
  Week 24 | -1.48 (1.894) | -2.07 (2.126) | -1.80 (1.896)

ADVERSE EVENTS:
Time Frame: Up to Day 172
Arm/Group | OnabotulinumtoxinA 400 U | OnabotulinumtoxinA 200 U | Placebo
Serious Adverse Events (participants affected / at risk) | 6/44 | 4/43 | 6/89
Other Adverse Events (participants affected / at risk) | 9/44 | 15/43 | 26/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA 400 U (N=44) | OnabotulinumtoxinA 200 U (N=43) | Placebo (N=89)
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA 400 U (N=44) | OnabotulinumtoxinA 200 U (N=43) | Placebo (N=89)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Hypertension (Vascular disorders) | 1 | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 2 | 8
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.